CLINICAL TRIAL: NCT00633451
Title: Randomized Clinical Trial of Rehabilitation for Subacromial Impingement Syndrome: A Comparison of Manual Therapy + Exercise to Exercise Only
Brief Title: Randomized Clinical Trial of Rehabilitation for Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Proaxis Therapy (Industry)
Collaborators: Virginia Commonwealth University (Other); Arcadia University (Other); National Athletic Trainers' Association Research & Education Foundation (NATA Foundation) (Other)
Responsible Party: Principal Investigator, Chuck Thigpen, Clinical Research Scientist, Proaxis Therapy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-173
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Shoulder Impingement Syndrome
Keywords: shoulder pain; shoulder impingement syndrome; manual therapy; rehabilitation
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Musculoskeletal Manipulations; Exercise; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Manual Therapy + Exercise
  Interventions: Other: Manual Therapy and Exercise
- 2 (Active Comparator): Exercise Only
  Interventions: Other: Exercise Only

INTERVENTIONS:
Other: Manual Therapy and Exercise — Manual therapy to the thoracic spine and shoulder, and therapeutic exercise to the shoulder and spine applied in a prescribed progression of therapeutic exercise aimed at improving shoulder function.
  Other Names: Manual Therapy and Therapeutic Exercise
  Arms: 1
Other: Exercise Only — A prescribed progression of therapeutic exercise for the shoulder and spine aimed at improving shoulder function
  Other Names: Therapeutic Exercise
  Arms: 2

SUMMARY:
The purpose of this randomized double-blind clinical trial is to determine the effectiveness of manual therapy for patients with subacromial impingement syndrome of the shoulder. We hypothesize that a combination of therapeutic exercise and manual therapy to the shoulder and spine will be more effective in reducing pain and shoulder disability at short-term (6 wk) and long-term (3, 6, 12 months) as compared to therapeutic exercise only.

DETAILED DESCRIPTION:
Subacromial impingement syndrome (SAIS) is a frequent cause of shoulder pain. Clinical trials investigating the effectiveness of manual therapy have demonstrated improvements in outcomes when manual therapy has been added to a program of therapeutic exercise. However, the these clinical trials (3) have significant limitations and generalizability. Two of the three 3 trials had a small number of subjects (14 & 22 subjects) and all 3 trials had only short term follow up (<12 weeks) and used non-validated self report outcome measures. These limitations reduce the confidence with which clinicians can apply these results to the patients they treat with SAIS. Clear evidence is needed to justify the cost and clinician time required to perform manual therapy in the delivery of patient care. Therefore, the purpose of this randomized clinical trial is to examine the short-term and long-term effectiveness of manual therapy in addition to therapeutic exercise as compared to therapeutic exercise only in patients diagnosed with SAIS.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms associated with athletic activity (35% of patients)
* Diagnosis of shoulder impingement syndrome as evidence by all 3 criteria:

  1. Reproduction of symptoms with impingement test: either Hawkins- Kennedy or Neer Test
  2. Pain during active shoulder elevation at or above 60 degrees
  3. Weakness of rotator cuff or pain during the Empty Can test or during resisted shoulder external rotation
* Shoulder disability: 25/100 (0 = no disability)
* Able to understand written and spoken

Exclusion Criteria:

* Severe pain; pain is > 7/10 on NPRS (0 = no pain)
* Shoulder surgery on affected shoulder
* Traumatic shoulder dislocation within the past 3 months
* Previous rehabilitation for this episode of shoulder pain
* Reproduction of shoulder pain with active or passive cervical motion
* Systemic inflammatory joint disease
* Global loss of passive shoulder ROM, indicative of adhesive capsulitis
* Full-thickness rotator cuff tear, as evidenced by any one of the following:

  1. Markedly reduced shoulder external rotation strength
  2. Drop arm test
  3. External rotation lag sign
  4. Lift off test
  5. Positive findings on MRI or ultrasonography

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Shoulder disability and pain | 6 weeks and 3, 6,12 months

SECONDARY OUTCOMES:
Patient satisfaction Quality of life (SF-36) Additional healthcare utilization and medication | 6 weeks, and 3, 6, 12 months
Patient perceived global rating of effect | 6 weeks and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Thigpen, PhD, PT, ATC, Principal Investigator — University of North Florida; Lori A Michener, PhD, PT, ATC, Principal Investigator — Virginia Commonwealth University; Phil McClure, PhD, PT, Principal Investigator — Arcadia University; Angela R Tate, PhD, PT, Study Director — Arcadia University
Locations (1):
- Proaxis Therapy, Greenville, South Carolina, United States

REFERENCES:
- See also: Related Info — http://www.proaxistherapy.com